CLINICAL TRIAL: NCT04252014
Title: Optimizing Hookah Tobacco Public Education Messages to Reduce Young Adult Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000277; R01CA229082 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-07

CONDITIONS: Hookah Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: The intervention consists of brief hookah tobacco public education messages delivered online through 4 brief study communications. Messages will communicate about the risks of hookah tobacco use in the following theme areas: 1) Health Harms; 2) Addictiveness; 3) Social Use; 4) Flavorings. The order of message themes delivered in each study communication will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Tobacco Messages (No Intervention): Participants in the control group will receive messages about health topics unrelated to tobacco use (e.g., sun safety). Messages will be delivered online through 4 brief study communications.
- Hookah Tobacco Messages (Experimental): Participants in the hookah tobacco messaging group will receive hookah tobacco public education messages delivered online through 4 brief study communications. Messages will communicate about the risks of hookah tobacco use in the following theme areas: 1) Health Harms; 2) Addictiveness; 3) Social Use; 4) Flavorings. The order of message themes delivered in each study communication will be randomized.
  Interventions: Behavioral: Hookah tobacco messages

INTERVENTIONS:
Behavioral: Hookah tobacco messages — Messages communicating the risks of hookah tobacco use in 4 thematic areas: health harms, addictiveness, social use, flavorings.
  Arms: Hookah Tobacco Messages

SUMMARY:
This is a 2-arm randomized controlled trial to test the effects of hookah tobacco public education messages among young adults who are susceptible non-users of hookah tobacco and those who are current hookah tobacco users. The primary outcomes are hookah tobacco use behavior (initiation among baseline susceptible non-users, frequency of use and cessation among baseline current users) at 6-month follow-up. Secondary outcomes are curiosity to use hookah tobacco (susceptible non-users) and motivation to quit using hookah tobacco (current hookah users) measured at 6-month follow-up. These outcomes will also be measured at 2- and 4-month follow-up time points.

DETAILED DESCRIPTION:
This is a 2-arm randomized controlled trial to test the effects of hookah tobacco public education messages among young adults who are susceptible non-users of hookah tobacco and current hookah tobacco users. Primary outcomes of hookah use behavior will be measured at the 6-month follow-up assessment. Secondary outcomes include curiosity to use hookah tobacco among susceptible non-users and motivation to quit using hookah tobacco among current users. All outcomes are also assessed at 2- and 4-month follow-up time points. All trial participants will be recruited from a US national consumer research panel. Eligible participants will be 1) young adults ages 18 to 30 (inclusive); 2) who have never used hookah tobacco but are deemed susceptible or report hookah tobacco use at least once within the past month; and 3) are enrolled members of the partnering consumer research panel. Panel members will be contacted via email with a brief description of the study and a link to an eligibility screener and online informed consent form. Eligible participants will complete a secure online baseline assessment of demographic characteristics, tobacco use history, and measures of hookah tobacco use behavior, beliefs, attitudes, and perceptions. After completing a baseline, participants will be randomly assigned in approximately equal numbers to one of two arms: 1) hookah tobacco messaging arm; 2) control arm. Through 4 brief study communications delivered approximately weekly, participants will receive study messages to which they are randomized and will complete brief self-report measures online on their responses to the messages. For the hookah tobacco messaging arm, communications will consist of study messages conveying risks of hookah tobacco use with random assignment of the order of messages with each exposure. In response to each message, participants will complete measures of message response and hookah-related beliefs, attitudes, and perceptions. Participants in the control condition will receive study communications with brief messages about health behaviors unrelated to tobacco (e.g., sun protection) and will complete the same measures. Hookah tobacco use behaviors, intentions and curiosity to use hookah tobacco (non-users), motivation to quit (current users), and hypothesized mediators will be assessed 2-, 4-, and 6-months after the message exposure period with the primary outcomes captured at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 30
* Smoked hookah tobacco within the past 30 days, OR never smoked hookah tobacco and deemed susceptible to using hookah tobacco based on answers to screening questions
* Member of partnering consumer research panel conducting the study

Exclusion Criteria:

* Age less than 18 or greater than 30
* Has not smoked hookah tobacco in the past 30 days OR has never smoked hookah tobacco and is not susceptible
* Not a member of partnering consumer research panel conducting the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 830 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, PhD, MPH, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie study results will be made available upon request by researchers after completion of the study and publication of primary findings.
Supporting Information: Study Protocol
Time Frame: After completion of the study and publication of the primary findings, for a period of up to 2 years.
Access Criteria: Investigators whose proposed use of the data have been approved by an independent review committee (i.e., IRB) for this purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Started | 414 | 416
Completed | 325 | 332
Not Completed | 89 | 84

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages | Total
Number analyzed (Participants) | 414 | 416 | 830
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (3.2) | 25.5 (3.1) | 25.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 247 | 506
  Male | 155 | 169 | 324
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 103 | 98 | 201
  Not Hispanic or Latino | 311 | 318 | 629
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 38 | 43 | 81
  Black | 129 | 113 | 242
  Multiple Races | 46 | 35 | 81
  Other Race(s) | 36 | 39 | 75
  White | 165 | 186 | 351
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 414 | 416 | 830

OUTCOME MEASURES:

1. Primary Outcome: Hookah Tobacco Initiation
Description: Hookah tobacco initiation among those who are susceptible non-users at baseline will be measured using a single valid survey question asking if participants have ever used hookah tobacco, even one or two puffs, at follow-up. The question asks if participants have ever smoked hookah tobacco based on a yes/no response. No hookah tobacco initiation is considered a better outcome. The outcome measure data reports those who responded "Yes" and are considered to have initiated hookah tobacco at the 6 month follow-up.
Time Frame: 6 months
Population: Participants who were susceptible never waterpipe smokers at baseline that were retained at the six month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 119 | 122
Participants | 11 | 5

2. Primary Outcome: Hookah Tobacco Use Frequency
Description: Hookah tobacco use frequency will be measured in baseline current hookah users with a single valid question asking on how many days they smoked hookah tobacco in the past 30 days. Baseline current hookah users who reported they quit were coded as smoking 0 of the past 30 days. Less frequent hookah use is considered a better outcome.
Time Frame: 6 months
Population: Participants who were current hookah smokers at baseline and retained to the 6 month follow-up. Some participants retained did not answer all outcomes questions.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 174 | 181
days | 2.52 (4.52) | 2.39 (4.51)

3. Primary Outcome: Hookah Tobacco Cessation
Description: Hookah tobacco cessation is measured using a single valid question adapted from the national Population Assessment of Tobacco and Health (PATH) survey asking participants who report they have not smoked hookah tobacco if they have stopped smoking hookah tobacco completely. The item asks if participants have completely stopped smoking hookah tobacco based on a yes/no response. Quitting hookah tobacco use (i.e., a response of "yes") is considered a better outcome. The outcome measure data reports those who responded "Yes" and are considered to have stopped smoking hookah tobacco completely at the 6 month follow-up.
Time Frame: 6 months
Population: Participants who were current hookah tobacco smokers at baseline retained to the 6 month follow-up. Some participants retained did not answer all outcomes questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 180 | 182
Participants | 66 | 55

4. Secondary Outcome: Hookah Tobacco Curiosity
Description: Curiosity to use hookah tobacco will be measured with a single valid item with a 7-point response ranging from 1 (not at all curious) to 7 (very curious) among those who are baseline susceptible non-users. This item will be administered at all time points. Outcomes from the 6-month follow-up are reported. A lower value on the response is considered a better outcome (i.e., less curious in using hookah tobacco).
Time Frame: 6 months
Population: Participants who were susceptible never hookah smokers at baseline retained to the 6 month follow-up. Some participants retained did not answer all outcomes questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 108 | 117
units on a scale | 2.01 (1.49) | 1.90 (1.27)

5. Secondary Outcome: Motivation to Quit Smoking Hookah Tobacco
Description: Motivation to quit smoking hookah tobacco will be measured with a single valid item with a 7-point response ranging from 1 (not at all motivated) to 7 (very motivated) among those who are current hookah users. This item will be administered at all time points. A higher value on the response is considered a better outcome (i.e., more motivated to quit smoking hookah tobacco). Outcomes at the 6-month follow-up are reported.
Time Frame: 6 months
Population: Baseline current hookah smokers who were retained at 6 month follow-up and did not quit. Some participants retained did not answer all outcomes questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 113 | 125
units on a scale | 3.82 (2.16) | 4.02 (2.30)

6. Other Pre Specified Outcome: Perceived Harm
Description: Perceived harm of hookah tobacco is measured using 4 self-report items. One item assesses perceptions of how harmful hookah tobacco use is (range 1 much less harmful than cigarettes to 5 much more harmful than cigarettes). Another item assesses how likely harms are to occur (range 1 no chance to 7 certain to happen). Another item assesses perceived harms of social hookah tobacco smoking in settings such as bars, cafes, and lounges (range 1 strongly disagree to 5 strongly agree). Another item assesses perceived harms of flavored hookah tobacco compared with unflavored hookah tobacco (range 1 strongly disagree to 5 strongly agree). For all 4 items, higher scores are considered better outcomes. The items are administered at 2-month, 4-month, and 6-month follow-up. Outcomes reported at 6-month follow-up reflect the sum of responses to the 4 items. The sum ranges from 4 (min) to 22 (max) with higher values considered better outcomes.
Time Frame: 6 months
Population: Participants at baseline who were retained to the 6 month follow up. Some participants retained did not answer all outcomes questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 324 | 329
units on a scale | 11.79 (2.42) | 11.85 (2.61)

7. Other Pre Specified Outcome: Perceived Addictiveness
Description: Perceived addictiveness of hookah tobacco is measured using 2 valid self-report items (Mays, Tercyak, & Lipkus 2016). The items assess perceptions of how addictive hookah tobacco smoking is on a 5 point response (1= much less addictive than cigarettes, 5 = much more addictive than cigarettes) and how likely one is to become addicted to hookah tobacco on a 7 point response(1 = no chance, 7 = certain to happen). Greater perceived addictiveness and perceived likelihood of addictiveness (higher values) are considered better outcomes. The items are administered at 2-month, 4-month, and 6-month follow-up. Outcomes reported are for the 6 month follow up timepoint and represent the sum of responses to the two items. The sum ranges from 2 (min) to 12 (max) with higher values considered better outcomes.
Time Frame: 6 months
Population: Participants at baseline who were retained to the 6 month follow-up. Some participants retained did not answer all outcomes questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 322 | 327
units on a scale | 6.81 (2.13) | 6.98 (2.30)

8. Other Pre Specified Outcome: Worry About Harm
Description: Worry about the harms of hookah tobacco is measured using a single valid self-report questionnaire item (Mays, Tercyak, & Lipkus 2016). The item assesses how much participants worry about the risks of hookah tobacco (1 = Not at all, 7 = Very much). Greater worry about harm is considered a better outcome. The items are administered at 2-month, 4-month, and 6-month follow-up.
Time Frame: 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 324 | 328
units on a scale | 4.29 (1.92) | 4.25 (2.04)

9. Other Pre Specified Outcome: Worry About Addictiveness
Description: Worry about the addictiveness of hookah tobacco is measured using a single valid self-report questionnaire item (Mays, Tercyak, & Lipkus 2016). The item assesses how much participants worry about becoming addicted to hookah tobacco (1 = Not at all, 7 = very much). Higher values indicate greater worry about addictiveness and are considered a better outcome. The items are administered at 2-month, 4-month, and 6-month follow-up.
Time Frame: 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
Number analyzed (Participants) | 324 | 330
units on a scale | 3.83 (2.00) | 3.87 (2.08)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Non-Tobacco Messages | Hookah Tobacco Messages
All-Cause Mortality (participants affected / at risk) | 0/414 | 0/416
Serious Adverse Events (participants affected / at risk) | 0/414 | 0/416
Other Adverse Events (participants affected / at risk) | 0/414 | 0/416

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04252014/Prot_SAP_000.pdf